CLINICAL TRIAL: NCT01156480
Title: Anti-inflammatory Treatment at the Onset of NEC in Preterm Infants- a Pilot Study
Brief Title: Anti-inflammatory Treatment at the Onset of Necrotizing Enterocolitis (NEC) in Preterm Infants
Acronym: steroids/NEC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Endeavor Health (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, Brandy Frost, Clinician Educator and Attending Neonatologist, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH09-196
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Necrotizing Enterocolitis
Keywords: necrotizing enterocolitis; NEC; premature; hydrocortisone; steroids; anti-inflammatory
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hydrocortisone (Experimental): Subjects in hydrocortisone group will receive 3mg/kg/day divided every 8 hours via intravenous (IV) route for 3 days, followed by 2mg/kg/day divided every 8 hours IV for 1 day, followed by 1.5mg/kg/day divided every 8 hours IV for 1 day, followed by 1mg/kg/day divided every 12 hours for 1 day, followed by 0.5mg/kg/day in single dose for one day. Subjects in placebo group will receive equal volume of placebo on the same dosing schedule. The first dose of study drug will be given within 6 hours of diagnosis of NEC, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
  Interventions: Drug: hydrocortisone
- Placebo (Placebo Comparator): Subjects in placebo group will receive equal volume of placebo (as compared to hydrocortisone arm) on the same dosing schedule. The first dose of study drug will be given within 6 hours of diagnosis of NEC, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: hydrocortisone — Subjects in hydrocortisone group will receive 3mg/kg/day divided every 8 hours via IV route for 3 days, followed by 2mg/kg/day divided every 8 hours IV for 1 day, followed by 1.5mg/kg/day divided every 8 hours IV for 1 day, followed by 1mg/kg/day divided every 12 hours for 1 day, followed by 0.5mg/kg/day in single dose for one day. The first dose of study drug will be given within 6 hours of diagnosis of NEC, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
  Arms: hydrocortisone
Drug: placebo — Subjects in placebo group will receive a volume of placebo equal to the hydrocortisone group, on the same dosing schedule, with doses given every 8 hours via IV route for 3 days, followed by placebo every 8 hours IV for 1 day, followed by placebo every 8 hours IV for 1 day, followed by placebo every 12 hours for 1 day, followed by placebo in single dose for one day. The first dose of study drug will be given within 6 hours of diagnosis of NEC, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
  Arms: Placebo

SUMMARY:
Despite modern medical advances, necrotizing enterocolitis (NEC) remains a significant problem in neonatal intensive care units (ICUs). Although research has shown NEC to be an inflammatory necrosis of the bowels, to date no study has examined the effect of anti-inflammatory therapy on this dreaded disease once it is diagnosed. The investigators propose a multi-center, randomized, placebo-controlled, double-blinded pilot study to examine the effect of hydrocortisone in infants diagnosed with stages II and III NEC. The investigators will follow C-reactive protein (CRP) levels as a marker of systemic inflammation for the primary outcome in this study.

DETAILED DESCRIPTION:
Given the extensive inflammatory response inherent to NEC, anti-inflammatory treatment may be of benefit, to both reduce inflammation and as a potential therapy to improve outcome. To date, there is no specific therapy for NEC that has been found to improve outcome, but corticosteroids have yet to be investigated in that capacity. Therefore, we propose to examine the effect of hydrocortisone for treatment of NEC in a randomized, blinded, placebo-controlled pilot study, focusing on a primary outcome of C-reactive protein levels at 3 and 7 days of therapy as a measure of inflammation. In addition, we will follow several secondary outcome measures to determine the possibility of improved outcome in those infants assigned to hydrocortisone.

The investigators hypothesize that infants diagnosed with NEC who receive hydrocortisone will have significantly lower C-reactive protein levels at 3 and 7 days of treatment versus infants who receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Infant born at gestational age less than 34 weeks
* Birth weight less than 2500 grams
* Diagnosis of stage II or III NEC made by attending neonatologist, neonatology fellow, or pediatric hospitalist
* Legally authorized representative is able to provide written informed consent prior to the performance of an protocol-specified evaluations or procedures
* Consent can be obtained and study drug can be administered within 6 hours of diagnosis

Exclusion Criteria:

* congenital gastrointestinal anomaly
* subject is already receiving parenteral steroid therapy or subject has received parenteral steroids within one week prior to study entry
* subject has received indomethacin therapy within 48 hours prior to being diagnosed with NEC

Ages: 0 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandy L Frost, MD, Principal Investigator — Endeavor Health
Locations (2):
- United States (2):
  - University of Chicago Comer Childrens Hospital, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrocortisone: hydrocortisone group will receive 3mg/kg/day divided every 8 hours via intravenous route for 3 days, then 2mg/kg/day divided every 8 hours IV for 1 day, then 1.5mg/kg/day divided every 8 hours IV for 1 day, then 1mg/kg/day divided every 12 hours for 1 day, then 0.5mg/kg/day in single dose for one day. Placebo group will receive equal volume of placebo on the same schedule. The first dose of study drug will be given within 6 hours of NEC diagnosis, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
Period: Overall Study
Arm/Group | Hydrocortisone | Placebo
Started | 0 | 2
Completed | 0 | 1
Not Completed | 0 | 1
Not completed — change in diagnosis | 0 | 1

BASELINE CHARACTERISTICS:
Population: premature neonates
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocortisone | Placebo | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 1 | 1
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 1 | 1
  Male |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: CRP Level
Description: C-reactive protein is a non-specific marker of inflammation, noted to be elevated in infants diagnosed with NEC.
Time Frame: 3 days
Population: This study was terminated due to low enrollment. We had a drop in our incidence of NEC, so there were very few eligible infants. One subject that was enrolled was soon thereafter thought NOT to have NEC, so that subject never received study drug.
Measure: Number; unit: mg/L
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
mg/L |  | 25.3

2. Primary Outcome: CRP Level
Description: C-reactive protein (CRP) is a non-specific measure of inflammation, usually elevated in infants diagnosed with NEC
Time Frame: 7 days
Population: as for outcome 1
Measure: Number; unit: mg/L
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
mg/L |  | 6.7

3. Secondary Outcome: Gastrointestinal (GI) Failure (Defined as Not Being on Full Enteral Feeds of 120kcal/kg/Day at 36 Weeks Corrected Age)
Description: GI failure
Time Frame: 36 weeks corrected gestational age
Population: The one enrolled infant did not have GI failure at 36 weeks CGA.
Measure: Count of Participants; unit: Participants
Groups:
- Hydrocortisone: Subjects in hydrocortisone group will receive 3mg/kg/day divided every 8 hours via intravenous (IV) route for 3 days, followed by 2mg/kg/day divided every 8 hours IV for 1 day, followed by 1.5mg/kg/day divided every 8 hours IV for 1 day, followed by 1mg/kg/day divided every 12 hours for 1 day, followed by 0.5mg/kg/day in single dose for one day. Subjects in placebo group will receive equal volume of placebo on the same dosing schedule. The first dose of study drug will be given within 6 hours of diagnosis of NEC, once informed consent is obtained, and subjects will continue to receive study drug until all doses have been given (total of 18 doses) or consent is withdrawn.
  hydrocortisone: Subjects in hydrocortisone group will receive 3mg/kg/day divided every 8 hours via IV route for 3 days, followed by 2mg/kg/day divided every 8 hours IV for 1 day, followed by 1.5mg/kg/day divided every 8 hours IV for 1 day, followed by 1mg/kg/day divided every 12 hours for 1 day, followed by 0.5mg/k
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 0

4. Secondary Outcome: Spontaneous Intestinal Perforation
Description: Whether or not infants had perforation.
Time Frame: at 36 weeks corrected gestational age
Population: Only 1 infant enrolled (placebo group)
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 0

5. Secondary Outcome: Need for Gastrointestinal Surgery
Description: Whether or not the infants required GI surgery by 36 weeks CGA
Time Frame: at 36 weeks corrected gestational age
Population: We only enrolled one subject (placebo group)
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 0

6. Secondary Outcome: Incidence of Sepsis
Description: Whether or not enrolled subjects had sepsis before 40 weeks CGA
Time Frame: at 40 weeks corrected gestational age
Population: We only enrolled one subject (placebo group). She did have fungal sepsis).
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 1

7. Secondary Outcome: Time on Parenteral Nutrition
Description: Total time on parenteral nutrition
Time Frame: at 40 weeks corrected gestational age
Population: Only one subject was enrolled (placebo group)
Measure: Number; unit: days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
days |  | 39

8. Secondary Outcome: Time to Full Enteral Feeds
Description: this will be assessed as the time needed to achieve full enteral feeds following the diagnosis of NEC. On average, it will be assessed at 40 weeks CGA, near the time of discharge, but there is a subset of infants who will not yet have achieved full enteral feeds at that time, so it may need to be assessed later than 40 weeks CGA
Time Frame: at 40 weeks corrected gestational age
Population: We only enrolled one subject into the placebo group.
Measure: Number; unit: days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
days |  | 35

9. Secondary Outcome: Length of Stay
Description: this will be assessed at the time of discharge, around 40 weeks CGA on average. A subset of infants may be discharged later than 40 weeks corrected gestational age (CGA), however, so these infants will need to have length of stay assessed later than 40 weeks CGA.
Time Frame: at 40 weeks corrected gestational age
Population: only one subject enrolled into placebo group
Measure: Number; unit: days
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
days |  | 141

10. Secondary Outcome: Growth Velocity
Description: Growth velocity after NEC diagnosis, in g/kg/day.
Time Frame: at 40 weeks CGA
Population: We only enrolled one subject into the placebo group.
Measure: Number; unit: grams/kg/d
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
grams/kg/d |  | 14.4

11. Secondary Outcome: Mortality
Time Frame: at 40 weeks corrected gestational age
Population: Only one subject was enrolled into the placebo group.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrocortisone | Placebo
Number analyzed (Participants) | 0 | 1
Participants |  | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: This study was terminated due to low enrollment. The one enrolled infant was later thought not to have NEC. There was no data to analyze.
Arm/Group | Hydrocortisone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
This study was terminated due to low enrollment. We had a drop in our incidence of NEC, so there were very few eligible infants. One subject that was enrolled was soon thereafter thought NOT to have NEC, so that subject never received study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes